CLINICAL TRIAL: NCT07211568
Title: Effect of Pancreatic Enzyme Replacement Therapy on Nutrition in Acute Pancreatitis: A Multicenter Double Blinded Randomised Placebo Controlled Trial.
Brief Title: PERT in Acute Necrotizing Pancreatitis
Acronym: PERT-ANP
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANP-PERT 1
Record Dates: First submitted 2025-09-19; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Acute Pancreatitis Necrotizing; Nutrition Assessment
Keywords: Nutrition in AP; PERT in AP; pancreatic exocrine insufficiency
MeSH Terms: conditions — Pancreatitis, Acute Necrotizing; Exocrine Pancreatic Insufficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PERT (Experimental): Enteric coated enzyme preparation containing: Lipase 25000U, Amylase 18000U, Protease 1000U. These medications are to be taken thrice daily with food (Breakfast, lunch and dinner)
  Interventions: Drug: Pancreatic Enzyme Replacement Therapy
- Placebo (Placebo Comparator): Similar appearing glucose capsules will be provided three times a day along with food (breakfast, lunch and dinner)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pancreatic Enzyme Replacement Therapy — Enteric coated pancreatic enzyme preparation
  Arms: PERT
Drug: Placebo — Similar appearing glucose capsules
  Arms: Placebo

SUMMARY:
In this multicenter, double blinded, placebo-controlled, 1:1 parallel group RCT, we propose to evaluate the impact of pancreatic exocrine replacement therapy on patients with acute necrotizing pancreatitis (ANP). We will include patients of 18-60yrs age and both genders with >50% pancreatic parenchymal necrosis and >10% loss of body weight.

The primary outcome measure is change in BMI at 3 months after enrolment. The intervention will include pancreatic enzyme consisting of 25000 IU of lipase and similar appearing placebo.

DETAILED DESCRIPTION:
Acute pancreatitis (AP), an inflammatory disorder of the pancreas, is mild and self-limiting in most patients. Around 10-20% of AP patients develop acute necrotizing pancreatitis (ANP) which is characterized by destruction of both pancreatic and peripancreatic tissue and is associated with high rate of morbidity and mortality due to both local and systemic complications1,2,3.

Early recognition and close monitoring of affected patients is crucial. Treatment consists of goal-directed intravenous fluid resuscitation, pain control, and enteral nutrition as early as possible. While sterile necrosis might resolve with above conservative measures, infected necrosis requires antibiotics and further interventions such as percutaneous drainage, minimally invasive surgeries, and endoscopic necrosectomy4.

In ANP patients there is direct destruction of acinar tissue that results in pancreatic exocrine insufficiency (PEI). In PEI there is insufficient secretion of pancreatic enzymes that causes inadequate nutrient digestion and absorption resulting in weight loss, malnutrition, metabolic bone disease and fat-soluble vitamins and mineral deficiencies5. The risk of PEI after ANP is about 25% over 3 years6. According to two meta-analysis5,7, PEI was found to be more prevalent during the index AP episode and it remained persistent in about half of the study population at follow-ups. They also reported that the risk of developing PEI is more in those with alcoholic etiology and severe and necrotizing pancreatitis.

Hence, management of PEI following ANP is important to improve nutritional status and quality of life. Pancreatic enzyme replacement therapy (PERT) is the mainstay of treatment for PEI. While the use of PERT is well-established in chronic pancreatitis, its efficacy in patients with ANP is still unclear. Hence, in this study, we aim to provide insights into the potential benefits of enzyme supplementation in patients with ANP by evaluating nutritional status, clinical outcomes, and quality of life.

This is a multicenter, double blinded, placebo-controlled, 1:1 parallel group RCT, we propose to evaluate the impact of pancreatic exocrine replacement therapy on patients with acute necrotizing pancreatitis (ANP). We will include patients of 18-60yrs age and both genders with >50% pancreatic parenchymal necrosis and >10% loss of body weight.

The primary outcome measure is change in BMI at 3 months after enrolment. The intervention will include pancreatic enzyme consisting of 25000 IU of lipase and similar appearing placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with AP according to the Revised Atlanta Classification diagnostic criteria
* Index episode of acute pancreatitis with at least 50% pancreatic parenchymal necrosis and greater than at least 10% loss of pre pancreatitis body weight at the time of screening
* Within 28 days of onset of disease
* Age 18-60 years
* Both genders

Exclusion Criteria:

* Underlying chronic pancreatitis
* Recurrent acute pancreatitis
* Pancreatic cancer
* Patients being discharged with NJ tubes
* Pregnancy and lactation
* Inability to give informed consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 188 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in Body Mass Index (BMI) | 3 months
  BMI will be measured at baseline and again at 3 months follow-up, with the difference between the two time points used to assess the effect of the intervention on patients' weight status.

SECONDARY OUTCOMES:
1. Change in Quality of Life | 3 months
  Quality of life will be assessed by the Short Form (SF)-36 tool. The lowest score in this tool is 0 and the highest score is 100, a higher score indicating better quality of life.
Change in pancreatic exocrine function | 3 months
  Exocrine function will be assessed by the Fecal elastase test.
Change in nutritional status: Anthropometry | 3 months
  Skin fold thickness over the triceps muscle at the mid arm level.
Change in nutritional status: Anthropometry | 3 months
  Mid-arm circumference
Change in nutritional status: Biochemical assessment | 3 months
  Serum prealbumin levels (gm/dL)
Change in nutritional status: Biochemical assessment | 3 months
  Serum vitamin D levels
Change in nutritional status: Biochemical assessment | 3 months
  Serum vitamin B12 levels
Change in the endocrine status | 3 months
  HbA1c and C-peptide
Change in patient's impression of change after treatment | 3 months
  This will be evaluated using the Patient's Global Impression of Change (PGIC). The score ranges from 1-7, with a score of 1 indicating very much improved and 7 indicating very much worse.
Readmission after onset of treatment | 3 months
  Readmission to hospital

CONTACTS AND LOCATIONS:
Overall Officials: Rupjyoti Talukdar, MD, Study Director — Asian Institute of Gastroenterology

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Huang W, de la Iglesia-Garcia D, Baston-Rey I, Calvino-Suarez C, Larino-Noia J, Iglesias-Garcia J, Shi N, Zhang X, Cai W, Deng L, Moore D, Singh VK, Xia Q, Windsor JA, Dominguez-Munoz JE, Sutton R. Exocrine Pancreatic Insufficiency Following Acute Pancreatitis: Systematic Review and Meta-Analysis. Dig Dis Sci. 2019 Jul;64(7):1985-2005. doi: 10.1007/s10620-019-05568-9. Epub 2019 Jun 4. PMID 31161524
- [Background] Umapathy C, Raina A, Saligram S, Tang G, Papachristou GI, Rabinovitz M, Chennat J, Zeh H, Zureikat AH, Hogg ME, Lee KK, Saul MI, Whitcomb DC, Slivka A, Yadav D. Natural History After Acute Necrotizing Pancreatitis: a Large US Tertiary Care Experience. J Gastrointest Surg. 2016 Nov;20(11):1844-1853. doi: 10.1007/s11605-016-3264-2. Epub 2016 Sep 12. PMID 27619808
- [Background] Lee PJ, Papachristou GI. New insights into acute pancreatitis. Nat Rev Gastroenterol Hepatol. 2019 Aug;16(8):479-496. doi: 10.1038/s41575-019-0158-2. PMID 31138897
- [Background] Wang GJ, Gao CF, Wei D, Wang C, Ding SQ. Acute pancreatitis: etiology and common pathogenesis. World J Gastroenterol. 2009 Mar 28;15(12):1427-30. doi: 10.3748/wjg.15.1427. PMID 19322914
- [Background] Banks PA, Bollen TL, Dervenis C, Gooszen HG, Johnson CD, Sarr MG, Tsiotos GG, Vege SS; Acute Pancreatitis Classification Working Group. Classification of acute pancreatitis--2012: revision of the Atlanta classification and definitions by international consensus. Gut. 2013 Jan;62(1):102-11. doi: 10.1136/gutjnl-2012-302779. Epub 2012 Oct 25. PMID 23100216